CLINICAL TRIAL: NCT04199624
Title: Assessment of Gastric pH Changes Induced by Ascorbic Acid Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Hala Fadda (Unknown); Butler University (Unknown)
Responsible Party: Principal Investigator, John M. Wo, Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2006413011
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hypochlorhydria
MeSH Terms: conditions — Achlorhydria | interventions — Omeprazole; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: omeprazole and ascorbic acid (Experimental)
  Interventions: Drug: Omeprazole 20mg; Dietary Supplement: Vitamin C

INTERVENTIONS:
Drug: Omeprazole 20mg — Omeprazole twice daily x 5 days
Dietary Supplement: Vitamin C — Ascorbic acid x 1 on day 5

SUMMARY:
This study evaluates the use of ascorbic acid, vitamin C, to temporary reduce gastric pH in individuals with omeprazole induced hypochlorhydria. All participants will receive ascorbic acid tablets to measure the change in gastric pH.

DETAILED DESCRIPTION:
Elevation of gastric pH in patients with hypochlorhydria can reduce the solubility of weakly basic drugs. This may lead to poor and unpredictable systemic exposure for poorly soluble drugs. For example, extent of absorption of the kinase inhibitors, dasatinib (Sprycel) and erlotinib (Tarceva), is reduced by up to 61% and 46% respectively in patients on acid-reducing agents (ARAs). This pilot study is to evaluate the use of ascorbic acid, vitamin C, to temporary reduce gastric pH in individuals with omeprazole induced hypochlorhdyria. Using pH/impedance testing, we are seeking to determine the magnitude and duration of pH change upon administration of 1000 mg of ascorbic acid in healthy subjects with proton-pump inhibitor induced hypochlorhydria. The results from this study will be used to evaluate the use of ascorbic acid as a drug-drug interaction mitigation strategy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, young males age 18-30 years with no prior history of gastrointestinal disease or symptoms.

Exclusion Criteria:

* Hypochlorhydria (baseline use antacids, antisecretory medications, or surface agents including proton-pump inhibitors, H2 blockers, or sucralfate).
* Current or previous history of gastrointestinal disease including gastroesophageal reflux disease, Barrett's esophagus, peptic ulcer disease, dyspepsia, gastroparesis, bacterial overgrowth, microscopic colitis, gastric intestinal metaplasia or metaplastic atrophic gastritis, gastric neuroendocrine tumors, helicobacter pylori infection, inflammatory bowel disease (Crohn's disease or ulcerative colitis), celiac disease, visceral cancer, chronic infectious disease, immunodeficiency, uncontrolled thyroid disease, history of liver disease).
* History of gastric bypass or other abdominal surgeries excluding cholecystectomy or appendectomy > 6 months prior to study initiation.
* Radiation therapy to the abdomen.
* Pregnant females.
* Ingestion of any prescription, over-the-counter, or herbal medications which may affect study interpretation.
* Currently a smoker
* Antibiotic use within the last 3 months

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological males
Enrollment: 11 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Change in gastric pH and duration of gastric pH \status | From time of inpatient appointment to thirteen months after that time point.
  Gastric pH measurements will be continuously monitored throughout the study using a catheter-based pH monitoring system. Gastric pH versus time data will be collected for five hours.

SECONDARY OUTCOMES:
Intestinal microbiome profile, intestinal metabolomic profile | From time of initial stool drop-off to thirteen months after that time point.
  To explore the correlation between physiologic responses in gastric pH with features of the intestinal microbiome and microbial metabolites (e.g. metabolome).

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No